# STUDY INFORMED CONSENT

Visual Attention to Text and Pictorial Food Labels: An Eye Tracking Experiment

NCT number NCT05958888 Document Date 05/23/2023 University of North Carolina at Chapel Hill Consent to Participate in a Research Study Survey Adult Participants

Consent Form Version Date: May 23, 2023

**IRB Study #** 23-0659

**Title of Study**: Food Perceptions Study **Principal Investigator**: Marissa Hall

Principal Investigator Department: Health Behavior
Principal Investigator Phone number: +1 (919) 966-0233
Principal Investigator Email Address: mghall@unc.edu
Funding Source and/or Sponsor: National Institutes of Health

Study Contact Telephone Number: +1 (919) 960-1662

Study Contact Email: storestudy@unc.edu

## **Concise Summary**

The purpose of this research study is to understand responses to different labels on food products. You are being asked to take part in a research study because you are an adult (age 18 or older) who identifies as Hispanic or Latino.

After consenting to take part in this study, you will visit our office in Carrboro, North Carolina one time. During the in-person visit, you will participate in an online computer activity that involves viewing different images. You'll then take a brief survey about your experience during the activity. The study visit will take 30-45 minutes. You will receive a \$40 incentive for your participation in this study.

Research is designed to benefit society by gaining new knowledge. You will not benefit personally from being in this research study. While we do not expect any risks to you during this study, one potential risk is loss of confidentiality. The study team will take steps to keep your information safe and private.

#### What are some general things you should know about research studies?

You are being asked to take part in a research study. To join the study is voluntary. You may choose not to participate, or you may withdraw your consent to be in the study, for any reason, without penalty.

Research studies are designed to obtain new knowledge. This new information may help people in the future. You may not receive any direct benefit from being in the research study. There also may be risks to being in research studies.

Details about this study are discussed below. It is important that you understand this information so that you can make an informed choice about being in this research study.

You may keep a copy of this consent form or request one by emailing calliew@unc.edu. You should ask the researchers named above, or staff members who may assist them, any

questions you have about this study at any time.

## What is the purpose of this study?

The purpose of this research study is to understand responses to different labels on food products.

You are being asked to take part in a research study because you are an adult (age 18 or older) who identifies as Hispanic or Latino/a/é.

# Are there any reasons you should not be in this study?

You should not be in this study if you:

- are under age 18
- have glaucoma
- are blind
- have cataracts
- have permanently dilated pupils
- have eye implants (artificial lenses; contact lenses are okay)
- wear bifocals

#### How many people will take part in this study?

Approximately 75 people will take part in this study.

# How long will your part in this study last?

About 30-45 minutes.

#### What will happen if you take part in the study?

You will be asked to participate in an activity on a computer that involves viewing images and answering questions about those images.

#### What are the possible benefits from being in this study?

Research is designed to benefit society by gaining new knowledge. You will not benefit personally from being in this research study.

#### What are the possible risks or discomforts involved from being in this study?

One potential risk for being in this study loss of privacy resulting from accidental disclosure of responses to survey questions or of data collected on purchases. Not only are these risks small, but the risk of a rare accidental disclosure would also be small because we are not collecting sensitive information. There may be uncommon or previously unknown risks. You should report any problems to the researcher or study team.

#### How will information about you be protected?

Participants will not be identified in any report or publication about this study. We may use deidentified data from this study in future research without additional consent. We may make a deidentified dataset from this study available publicly when we publish the results. Although every effort will be made to keep research records private, there may be times when federal or state law requires the disclosure of such records, including personal information. This is very unlikely, but if disclosure is ever required, UNC-Chapel Hill will take steps allowable by law to protect the privacy of personal information. In some cases, your information in this research study could be reviewed by representatives of the University, research sponsors, or government agencies (for example, the FDA) for purposes such as quality control or safety. What is a Certificate of Confidentiality? This research is covered by a Certificate of Confidentiality. With this Certificate, the researchers may not disclose or use information, documents or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings in the United States, for example, if there is a court subpoena, unless you have consented for this use.

The Certificate cannot be used to refuse a request for information from personnel of a federal or state agency that is sponsoring the study for auditing or evaluation purposes or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA).

The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law, such as mandatory reporting requirements for child abuse or neglect, disabled adult abuse or neglect, communicable diseases, injuries caused by suspected criminal violence, cancer diagnosis or benign brain or central nervous system tumors or other mandatory reporting requirement under applicable law. The Certificate of Confidentiality will not be used if disclosure is for other scientific research, as allowed by federal regulations protecting research subjects or for any purpose you have consented to in this informed consent document.

You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

#### What if you want to stop before your part in the study is complete?

You can withdraw from this study at any time, without penalty. The investigators also have the right to stop your participation at any time. If you withdraw or are withdrawn from this study all data collected up until the point of withdrawal will be retained, however no additional information will be collected unless you provide additional written permission for further data collection at the time of your withdrawal.

## Will you receive anything for being in this study?

You will receive a \$40 incentive for participating in this study.

#### Will it cost you anything to be in this study?

You will need to provide transportation to the study site (in Carrboro, North Carolina). It will not cost you anything else to be in this study.

#### Who is sponsoring this study?

This research is funded by the National Institutes of Health. This means that the research team is being paid by the sponsor for doing the study. The researchers do not, however, have a direct financial interest with the sponsor or in the final results of the study.

## What if you have questions about this study?

You have the right to ask, and have answered, any questions you may have about this research. If you have questions about the study (including payments), complaints, concerns, or if a research-related injury occurs, you should contact the study team members listed on the first page of this form.

| IRB TEMPLATE Version 2.2 - 10/26/2020 - Do not alter t |
|--------------------------------------------------------|
|--------------------------------------------------------|

# What if you have questions about your rights as a research participant?

All research on human volunteers is reviewed by a committee that works to protect your rights and welfare. If you have questions or concerns about your rights as a research subject, or if you would like to obtain information or offer input, you may contact the Institutional Review Board at 919-966-3113 or by email to <a href="mailto:IRB">IRB</a> subjects@unc.edu.

**Note:** If you indicated that you were interested in hearing about future research studies, we will maintain your contact information indefinitely, separate from any other study data.

# **Subject's Agreement:**

| I have read the information provided above. I have asked all the voluntarily agree to continue to participate in this research study. | • |
|---|---|
| Signature of Research Subject | Date |
| Printed Name of Research Subject | |
| Signature of Research Team Member Obtaining Consent | Date |
| Printed Name of Research Team Member Obtaining Consent | |